CLINICAL TRIAL: NCT03145480
Title: Two-arm Phase II Trial Exploring the Use of the Targeted Agents Ibrutinib and Obinutuzumab for the Treatment of Patients With a Diagnosis of Richter's Transformation (RT) or Richter's Syndrome (RS)
Brief Title: Study of Ibrutinib & Obinutuzumab With/Without CHOP for Richter's Transformation or Richter's Syndrome Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decision to close study
Sponsor: Northwell Health (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-727
Record Dates: First submitted 2017-04-04; First posted 2017-05-09 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Richter Syndrome
Keywords: leukemia; richter
MeSH Terms: conditions — Leukemia | interventions — obinutuzumab; ibrutinib; VAP-cyclo protocol

STUDY DESIGN:
Intervention Model Description: parallel assignment based on fitness of participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fit arm (Experimental): ibrutinib and obinutuzumab in combination with the CHOP regimen
  Interventions: Drug: Obinutuzumab; Drug: Ibrutinib; Other: CHOP
- Frail arm (Experimental): ibrutinib and obinutuzumab
  Interventions: Drug: Obinutuzumab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Obinutuzumab — 100 mg on day 1 and 900 mg on day 2 Cycle 1, 1000 mg on day 8 and 15 of Cycle 1, and 1000 mg on day 1 of Cycles 2-6
  Other Names: gazyva
Drug: Ibrutinib — 560mg po daily
  Other Names: imbruvica
Other: CHOP — cyclophosphamide, doxorubicin, vincristine, and prednisone
  Other Names: CHOP Regimen
  Arms: Fit arm

SUMMARY:
This research study studies the combination of ibrutinib and obinutuzumab with or without the standard chemotherapy regimen of CHOP to see how well these drugs work in treating patients with a diagnosis of Richter's Transformation or Richter's Syndrome. The Bruton's Tyrosine Kinase (BTK) inhibitor, ibrutinib, may stop growth of cancer cells by blocking the signal needed for cell growth. The monoclonal antibody obinutuzumab may block cancer growth by targeting cells present in Richter's Transformation. Giving ibrutinib with obinutuzumab may be a better treatment for patients with Richter's Transformation. Depending on fitness, the patients may receive ibrutinib and obinutuzumab in combination with a regimen known as CHOP (C= cyclophosphamide, H= hydroxydaunorubicin (also called doxorubicin), O= oncovin (also called vincristine, and P= prednisolone or prednisone (corticosteroids).

ELIGIBILITY:
Inclusion Criteria:

* confirmed Richter's transformation in treatment naïve and previously treated chronic lymphocytic leukemia/small lymphocytic lymphoma patients
* may have had prior exposure to ibrutinib and other B-cell signaling receptor agents
* Adequate hematologic function
* Adequate liver and kidney function
* Willing and able to participate in all required evaluations and procedures in this study protocol
* Female subjects of childbearing potential must not be pregnant upon study entry
* Male and female subjects who agree to use highly effective methods of birth control

Exclusion Criteria:

* known allergy to any of medications
* chemotherapy taken within 21 days of study treatment
* targeted therapy within 10 days of study treatment
* BCR inhibitors within 24 hours of study treatment
* major surgery within 4 weeks of first dose of study treatment
* women who are pregnant
* known infection with HIV or Hepatitis C
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Barrientos, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health/CLL Research and Treatment Program, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fit Arm | Frail Arm
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Participants were only randomized to the Fit arm, no participants were in the Frail arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fit Arm | Frail Arm | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Customized [Count of Participants; unit: Participants]
  >= 18 Years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR in subjects treated with combination of ibrutinib and obinutuzumab (with or without CHOP)
Time Frame: 6 months
Population: No data was collected for this outcome measure.
Arm/Group | Fit Arm | Frail Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Improved Hemoglobin and Platelet Counts.
Description: hematologic improvement
Time Frame: 6 months
Population: No data was collected for this outcome measure.
Arm/Group | Fit Arm | Frail Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: time to progression post treatment of condition
Time Frame: 6 months
Population: No participants were enrolled into the Frail Arm. No data was collected for the Frail Arm, there are no results to report. Data reported for the Fit Arm is estimated.
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Fit Arm | Frail Arm
Number analyzed (Participants) | 3 | 0
Months | 23.5 (1.9) |

4. Secondary Outcome: To Evaluate Patient-reported Outcome (PRO) of Health-related Quality of Life by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACiT-Fatigue)
Description: health-related quality of life using FACIT Fatigue Scale
Time Frame: 1 year
Population: No data was collected for this outcome measure.
Arm/Group | Fit Arm | Frail Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year and 3 months
Description: No subjects were randomized to the Frail Arm, therefore no subjects were at risk for Adverse Events in this arm.
Arm/Group | Fit Arm | Frail Arm
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fit Arm (N=3) | Frail Arm (N=0)
neutropenia (Blood and lymphatic system disorders) | 1 (1) | NA — Grade 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | NA — Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fit Arm (N=3) | Frail Arm (N=0)
peripheral neuropathy (Nervous system disorders) | 1 (1) | NA — Grade 1
constipation (Gastrointestinal disorders) | 1 (1) | NA — Grade 1
hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | NA — Grade 1
hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | NA — Grade 1
fatigue (General disorders) | 3 (3) | NA — Grade 2
Anemia (Blood and lymphatic system disorders) | 2 (2) | NA
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | NA
diarrhea (Gastrointestinal disorders) | 1 (1) | NA
Alkaline phosphatase elevated (Investigations) | 1 (1) | NA
ALT increased (Investigations) | 1 (1) | NA
AST increased (Investigations) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT03145480/Prot_SAP_000.pdf